CLINICAL TRIAL: NCT05771337
Title: Circular RNA and Chemerin in Blood of Breast Cancer Patients
Brief Title: Circular RNA and Chemerin in Breast Cancer Patient
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sandy Nashat Sorial Shokrey, demonstrator in biochemestry departement, Assiut University
Other Study IDs: biomarkers in breast cancer
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- breast cancer leasion
  Interventions: Diagnostic Test: blood sample
- benign breast lesion
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — blood sample

SUMMARY:
This study aimed to evaluate the role of serum chemerin as a biomarker of breast cancer.

and To investigate the diagnostic value of hsa_circ_0001785 (Circ-ELP3) and hsa_circ_100219 (Circ-FAF1) in serum samples of breast cancer patients to find out whether these circRNAs can utilize as a diagnostic and prognostic biomarker for human breast cancer assessment and make Correlation between serum chemerin levels , serum Circ-FAF1 , serum CircELP3 and classical tumor markers (CEA + CA15-3).

andTo elucidate if there is a difference between metastatic and non-metastatic cases as regard serum chemerin levels, serum Circ-FAF1 or Circ-ELP3.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women and despite advances in therapy over the past few decades, drug resistance, recurrence, metastasis and the heterogeneity of the cancer continue to be a problem in successful management of the diseases(Hong et al ,2019) .

Circular RNAs (CircRNAs) are single-stranded, covalently closed RNA molecules that are ubiquitous across species ranging from viruses to mammals(Zhou et al 3 .,2020). circRNAs can be divided into two categories including coding and noncoding circRNAs(Li et al., 2019) A new subtype of RNAs is circular RNAs, single-strand RNA molecules with less than 100 to more than 4,000 nucleotides (Lu et al., 2016) and a covalently closedloop structure. These molecules are produced through a backsplicing mechanism, in which the downstream 5'-end of the splice donor joins the upstream 3'-end splice acceptor and forms a product with a circular structure (wang et al., 2017).

Chemerin is a leukocyte chemoattractant widely expressed in many tissues and is known to recruit innate leukocytes.

Recently, more and more studies focus on the relationship between chemerin and cancers and found that chemerin acts an essential role in cancers.(Shin et al,2018) Chemerin expression is different depending on the tumor type (Zhang Y et al, 2013) the clinical significance of chemerin in breast cancer has been only reported by a very limited number of studies (EL Sagheer et al,2018).

ELIGIBILITY:
Inclusion Criteria:

* histopathological diagnosis of breast cancer

Exclusion Criteria:

* history of other types of cancers
* history of HIV
* history of any therapeutic interventions in form of chemo or hormonal therapy before specimen collection

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female with breast cancer
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
measure chemerin and Circular RNA in breast cancer patients | 2 years
  To elucidate if there is a difference between metastatic and non-metastatic cases as regard serum chemerin levels, serum Circ-FAF1 or Circ-ELP3.

REFERENCES:
- [Background] Song Y, Zhu X, Lin Z, Luo L, Wen D. The potential value of serum chemerin in patients with breast cancer. Sci Rep. 2021 Mar 22;11(1):6564. doi: 10.1038/s41598-021-85986-w. PMID 33753802
- [Background] Omid-Shafaat R, Moayeri H, Rahimi K, Menbari MN, Vahabzadeh Z, Hakhamaneshi MS, Nouri B, Ghaderi B, Abdi M. Serum Circ-FAF1/Circ-ELP3: A novel potential biomarker for breast cancer diagnosis. J Clin Lab Anal. 2021 Nov;35(11):e24008. doi: 10.1002/jcla.24008. Epub 2021 Sep 21. PMID 34545638